CLINICAL TRIAL: NCT02243098
Title: An Open-label, One-sequence Cross Over, Single Centre Trial, Investigating the Influence of Semaglutide on the Pharmacokinetics of Single Doses of Atorvastatin and Digoxin in Healthy Subjects
Brief Title: Investigating the Influence of Semaglutide on the Pharmacokinetics of Single Doses of Atorvastatin and Digoxin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NN9535-3818; 2013-001288-22 (EudraCT Number); U1111-1140-8551 (Other: WHO)
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide; Digoxin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Semaglutide (Experimental)
  Interventions: Drug: semaglutide; Drug: digoxin; Drug: atorvastatin

INTERVENTIONS:
Drug: semaglutide — Administered as a subcutaneous injection (s.c., under the skin). Initiated with weekly semaglutide dosing of 0.25 mg in the first 4 weeks, 0.5 mg the next 4 weeks, and 1.0 mg in the third 4 week period.
Drug: digoxin — Oral administration. Digoxin will be given as 2 single doses of 0.5 mg.
Drug: atorvastatin — Oral administration. Atorvastatin will be given as 2 single doses of 40 mg.

SUMMARY:
The trial is conducted in Europe. The aim of the trial is to investigate the influence of semaglutide on the pharmacokinetics (the exposure of the trial drug in the body) of single doses of atorvastatin and digoxin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, age between 18 and 55 years (both inclusive) at the time of signing informed consent
* Body mass index between 20.0 and 29.9 kg/m^2 (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method. Women of child-bearing potential must use an effective method of birth control throughout the trial including the 5 weeks follow-up period. Only highly effective methods of birth control are accepted (i.e. one that results in less than 1% per year failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine device), or sexual abstinence or vasectomised partner
* Any clinically significant disease history, in the opinion of the investigator, or systemic or organ disease including: cardiac, pulmonary, gastrointestinal, hepatic, neurologic, renal, genitourinary and endocrine, dermatologic or hematologic diseases
* Use of prescription or non-prescription systemic or topical medicinal products (including routine or non-routine vitamins or herbal supplements, but excluding paracetamol and contraceptives) within 3 weeks (or within 5 half-lives of the medicinal product, whichever is longest) prior to Visit 2 (first dose administration)
* History of drug/chemical substance abuse within 1 year from screening, or a positive result in the urine drug test
* History of alcohol abuse within 1 year from screening, or a positive result in the alcohol urine test, or consumption of more than 21 units (male)/14 units (female) of alcohol weekly (one unit of alcohol equals about 250 mL of beer or lager, one glass (120 mL) of wine, or 20 mL spirits)
* Smoking in the last 3 months prior to screening or a positive nicotine test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2015-04-07 (Actual); Study Completion 2015-04-07 (Actual)

PRIMARY OUTCOMES:
Area under the atorvastatin plasma concentration-time curve | From time 0 to 72 hours after a single dose
Area under the digoxin plasma concentration-time curve | From time 0 to 120 hours after a single dose

SECONDARY OUTCOMES:
Maximum observed atorvastatin plasma concentration | From time 0 to 72 hours after a single dose
Maximum observed digoxin plasma concentration | From time 0 to 120 hours after a single dose
Number of treatment emergent AEs (TEAEs) | From baseline (Visit 2, Day 1) to follow-up (Visit 12, 20 weeks after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Result] Hausner H, Derving Karsbol J, Holst AG, Jacobsen JB, Wagner FD, Golor G, Anderson TW. Effect of Semaglutide on the Pharmacokinetics of Metformin, Warfarin, Atorvastatin and Digoxin in Healthy Subjects. Clin Pharmacokinet. 2017 Nov;56(11):1391-1401. doi: 10.1007/s40262-017-0532-6. PMID 28349387
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com